CLINICAL TRIAL: NCT01543958
Title: Sevelamer Carbonate for Reducing Endotoxemia and Immune Activation: A Proof of Concept Study
Brief Title: Sevelamer for Reducing Endotoxemia and Immune Activation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5296; 1U01AI068636 (NIH)
Record Dates: First submitted 2012-02-29; First posted 2012-03-05 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-09

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — Sevelamer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sevelamer carbonate (Experimental): Patients will be administered two 800 mg tablets of Sevelamer carbonate orally three times a day for 8 weeks.
  Interventions: Drug: Sevelamer carbonate; Device: Sevelamer carbonate

INTERVENTIONS:
Drug: Sevelamer carbonate — Patients will be administered two 800 mg tablets of Sevelamer carbonate orally three times a day for 8 weeks.
  Other Names: Renvela
Device: Sevelamer carbonate
  Other Names: Renvela

SUMMARY:
HIV-infected people can have an increase in inflammation in their body organs, even after taking anti-HIV medicines.

Sevelamer carbonate is used to bind phosphate in dialysis patients. It can also bind endotoxin in the gut and lowers endotoxin levels in the blood of dialysis patients. Sevelamer carbonate decreases the inflammation endotoxin causes in dialysis patients.

A5296 is a phase II, single-arm study to evaluate the effect of 8 weeks of sevelamer carbonate administration on markers of microbial translocation and T-cell activation in the blood in chronically HIV-infected subjects not receiving ART.

DETAILED DESCRIPTION:
HIV-infected people can have an increase in inflammation in their body organs, even after taking anti-HIV medicines. Inflammation is a normal body reaction to any infection. However, if inflammation lasts a long time like in HIV infection, it may lead to complications, such as heart disease, cancer, liver disease, and problems with thinking. Also, HIV-infected people with high inflammation have lower CD4+ T-cell counts (cells that fight infection). Many HIV researchers are studying the harmful effects of this prolonged inflammation and possible ways to prevent these complications.

The increase in inflammation in HIV-infected people may be caused by HIV or by other factors such as parts of bacteria. These bacterial pieces, called endotoxins, do not cause harm in the intestine (gut). However, in HIV infection, there is damage to the gut that allows endotoxins to cross from the gut into the blood. These endotoxins then cause inflammation in the body. New research is focusing on strategies to reduce the levels of endotoxin as a way to decrease inflammation.

A drug called sevelamer carbonate is used to bind phosphate in dialysis patients. However, sevelamer carbonate also binds endotoxin in the gut and lowers endotoxin levels in the blood of dialysis patients. Sevelamer carbonate also decreases the inflammation endotoxin causes in dialysis patients. This study will see if sevelamer carbonate can have the same effects in HIV-infected patients.

A5296 is a phase II, single-arm study to evaluate the effect of 8 weeks of sevelamer carbonate administration on markers of microbial translocation as well as monocyte and T-cell activation in the blood in chronically HIV-infected subjects with CD4+ T-cell count ≥ 400 cells/mm3 not receiving ART. This study enrolled 40 subjects. To assess whether there is a persistent effect of study drug, subjects were observed for an additional 8 weeks off sevelamer carbonate and changes in biomarkers were monitored.

As A5296 is a phase II study of biologic activity, the primary and secondary analyses are as-treated, limited to subjects who have data for baseline and week 8 and who remain on study treatment through week 8. For any subject who initiated antiretroviral treatment (ART), analyses only included data collected prior to the time ART was started.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* No plans to initiate ART during the course of the proposed study.
* Screening CD4+ T-cell count ≥ 400 cells/mm3 performed in a laboratory that has a Clinical Laboratory Improvement Amendments (CLIA) certification or its equivalent.
* HIV-1 RNA >50 copies/mL within the last 180 days prior to entry.
* Screening serum phosphate > 2.6 mg/dL within 60 days prior to entry.
* Certain laboratory values, as detailed in section 4.1.6 of the protocol, obtained within 30 days prior to entry
* Female subjects of reproductive potential must have a negative serum or urine pregnancy test performed within 30 days prior to entry.
* Female subjects participating in sexual activity that could lead to pregnancy must agree to use at least one of the following forms of birth control for at least 30 days prior to study entry until the final study visit:

  * Condoms (male or female) with or without a spermicidal agent
  * Diaphragm or cervical cap with spermicide
  * Intrauterine device (IUD)
  * Hormone-based contraceptive
* Female subjects who are not of reproductive potential are eligible without requiring the use of a contraceptive.
* Confirmation of the availability of the stored pre-entry plasma and peripheral blood mononuclear cell (PBMC) samples for endotoxin, sCD14, and immune activation determinations, obtained from a fasting sample.
* Ability and willingness of subject to provide informed consent.
* No plans to use probiotics (defined as products that contain significant amounts of live microorganisms and are ingested for specific health benefits, e.g., yogurt with live and active cultures, Lactobacillus GG, Saccharomyces boulardii) during the study.

Exclusion Criteria:

* Known diagnosis of acute HIV infection within 180 days prior to study entry.
* Pregnant or breastfeeding.
* Use of any antiretroviral agent within 24 weeks prior to study entry.
* Use of systemic cancer chemotherapy or radiation therapy, immunosuppressive or immunomodulatory therapy (e.g., interferons, tumor necrosis factor antagonists, interleukins, systemic corticosteroids) within 24 weeks prior to study entry.

NOTE A: Use of inhaled steroids, nasal steroids, topical steroids, or the equivalent of 10 mg of prednisone or less per day or a less than 2-week course of oral steroids is not exclusionary.

NOTE B: A single course of 1% hydrocortisone cream applied up to 3 times a day to <10 square inches area for <2 weeks is permitted while on study. Use of all other topical steroids is excluded.

* Known allergy/sensitivity or any hypersensitivity to components of the study drug or its formulation.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Serious illness requiring systemic treatment and/or hospitalization within 60 days prior to study entry.
* Known cirrhosis or severe liver disease (e.g., ascites, encephalopathy, history of variceal bleeding).

NOTE: Potential subjects with chronic hepatitis B or C virus infection who do not have known cirrhosis or severe liver disease may participate in the study.

* Severe kidney disease (defined as estimated glomerular filtration rate [GFR] <30 mL/min/1.73m2) at screening.
* History of bowel obstruction or severe GI motility disorders including severe constipation.
* Severe dysphagia or swallowing disorders.
* Major GI tract surgery within 60 days prior to study entry.
* Intent to initiate or change the dose of lipid-lowering drugs during study. NOTE: Potential subjects on stable doses of lipid-lowering agents (defined as no change in preparation or dose within 90 days prior to study entry) are permitted and may be enrolled.
* Use of investigational therapies within 90 days prior to study entry unless permission was granted by the A5296 protocol chairs (see Study Management page).
* Currently receiving hepatitis C therapy or anticipation that such therapy will be started during the study.
* Use of probiotics, for more than 3 consecutive days within the 60 days prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-11; Primary Completion 2012-09 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Gandhi, MD, Study Chair — Massachusetts General Hospital ACTG CRS; Netanya Sandler, MD, Study Chair — National Institutes of Health (NIH)
Locations (15):
- United States (15):
  - Alabama Therapeutics CRS (5801), Birmingham, Alabama
  - UCLA CARE Center CRS (601), Los Angeles, California
  - Ucsf Aids Crs (801), San Francisco, California
  - Harbor-UCLA Med. Ctr. CRS (603), Torrance, California
  - University of Colorado Hospital CRS (6101), Aurora, Colorado
  - Univ. of Miami AIDS CRS (901), Miami, Florida
  - Northwestern University CRS (2701), Chicago, Illinois
  - Massachusetts General Hospital ACTG CRS (101), Boston, Massachusetts
  - Washington University CRS (2101), St Louis, Missouri
  - AIDS Care CRS (1108), Rochester, New York
  - Univ. of Rochester ACTG CRS (1101), Rochester, New York
  - Univ. of Cincinnati CRS (2401), Cincinnati, Ohio
  - Case CRS (2501), Cleveland, Ohio
  - Metro Health CRS (2503), Cleveland, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS (6201), Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Sandler NG, Zhang X, Bosch RJ, Funderburg NT, Choi AI, Robinson JK, Fine DM, Coombs RW, Jacobson JM, Landay AL, Douek DC, Tressler R, Read SW, Wilson CC, Deeks SG, Lederman MM, Gandhi RT; AIDS Clinical Trials Group A5296 Team. Sevelamer does not decrease lipopolysaccharide or soluble CD14 levels but decreases soluble tissue factor, low-density lipoprotein (LDL) cholesterol, and oxidized LDL cholesterol levels in individuals with untreated HIV infection. J Infect Dis. 2014 Nov 15;210(10):1549-54. doi: 10.1093/infdis/jiu305. Epub 2014 May 26. PMID 24864123

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A5296 accrual opened under protocol version 1.0 on 11/21/11, and the first subject was enrolled on 12/29/11. Accrual to the study closed on 8/1/12, with a total of 40 subjects enrolled from 15 sites within the US.
Period: Overall Study
Arm/Group | Sevelamer Carbonate
Started | 40
Completed | 36
Not Completed | 4
Not completed — Loss to follow-up | 3
Not completed — ART initiation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 1
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 44 [34 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 29
Race/Ethnicity, Customized [Number; unit: participants]
  White non-Hispanic | 10
  Black Non-Hispanic | 24
  Hispanic (regardless of Race) | 6
Region of Enrollment [Number; unit: participants]
  United States | 40
Log10 HIV-1 RNA [Median (Inter-Quartile Range); unit: copies/mL] | 3.58 [2.94 to 4.17]
CD4 count [Median (Inter-Quartile Range); unit: cells/mm^3] | 580 [494 to 716]

OUTCOME MEASURES:

1. Primary Outcome: Change in Endotoxin
Description: Change in LPS from baseline to week 8, where baseline value is the average of pre-entry and entry values.
Time Frame: baseline and Week 8
Population: This is an as-treated analysis, limited to 36 subjects who have data for baseline and week 8 and who remain on study treatment through week 8. All 36 subjects had valid data at both baseline and week 8 and were included in primary analysis.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 36
pg/mL | 0.20 [-4.06 to 5.81]
Statistical Analysis 1: Comparison: Sevelamer Carbonate; Test type: Superiority or Other; p = 0.87, Sign test — not adjusted for multiple comparisons; no other adjustment

2. Primary Outcome: Change in Soluble CD14 (sCD14)
Description: Change in soluble CD14 (sCD14) from baseline to week 8, where baseline value is the average of pre-entry and entry
Time Frame: baseline and week 8
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ug/mL
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 36
ug/mL | -0.02 [-0.18 to 0.06]
Statistical Analysis 1: Comparison: Sevelamer Carbonate; Test type: Superiority or Other; p = 0.62, Sign test — Not adjusted for multiple comparisons; no other adjustment

3. Secondary Outcome: Change in Endotoxin
Description: Change in endotoxin from baseline to week 4, where baseline value is the average of pre-entry and entry
Time Frame: baseline and week 4
Population: This is an as-treated analysis, limited to 36 subjects who have data for baseline and week 8 and who remain on study treatment through week 8. All 36 subjects had valid data at both baseline and week 4 and were included in this secondary analysis.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 36
pg/mL | 1.08 [-2.51 to 7.71]

4. Secondary Outcome: Change in Endotoxin
Description: Change in endotoxin from week 8 to week 16
Time Frame: week 8 and week 16
Population: This is an as-treated analysis, limited to 36 subjects who have data for baseline and week 8 and who remain on study treatment through week 8. Among these 36 subjects, 33 subjects with valid endpoint at both week 8 and week 16 were included in this secondary analysis.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 33
pg/mL | -2.39 [-8.04 to 2.65]

5. Secondary Outcome: Change in sCD14
Description: Change in sCD14 from baseline to week 4, where baseline value is the average of pre-entry and entry
Time Frame: baseline and week 4
Population: This is an as-treated analysis, limited to 36 subjects who have data for baseline and week 8 and who remain on study treatment through week 8. All 36 subjects have valid data at baseline and week 4 and were included in this secondary analysis.
Measure: Median (Inter-Quartile Range); unit: ug/mL
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 36
ug/mL | -0.09 [-0.23 to 0.11]

6. Secondary Outcome: Change in sCD14
Description: Change in sCD14 from week 8 to week 16
Time Frame: week 8 and week 16
Population: This is an as-treated analysis, limited to 36 subjects who have data for baseline and week 8 and who remain on study treatment through week 8. Among these 36 subjects, 34 subjects had valid data at both week 8 and week 16 and were included in this secondary analysis.
Measure: Median (Inter-Quartile Range); unit: ug/mL
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 34
ug/mL | 0.06 [-0.03 to 0.24]

7. Secondary Outcome: Change in CD4+ T-cell Activation
Description: Change from baseline to week 8 in CD4+ T-cell activation, defined as the %CD38+/HLA-DR+, where baseline value is the average of pre-entry and entry
Time Frame: baseline and week 8
Population: This is an as-treated analysis, limited to 36 subjects who have data for baseline and week 8 and who remain on study treatment through week 8. Among these 36 subjects, 33 subjects with valid data at baseline and week 8 were included in this secondary analysis.
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 33
percentage | 0.050 [-0.650 to 2.600]

8. Secondary Outcome: Change in CD4+ T-cell Activation
Description: Change from baseline to week 4 in CD4+ T-cell activation, defined as the %CD38+/HLA-DR+, where baseline value is the average of pre-entry and entry
Time Frame: baseline and week 4
Population: This is an as-treated analysis, limited to 36 subjects who have data for baseline and week 8 and who remain on study treatment through week 8. Among these 36 subjects, 35 subjects with valid data at baseline and week 4 were included in this secondary analysis.
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 35
percentage | 0.4 [-0.95 to 1.2]

9. Secondary Outcome: Change in CD4+ T-cell Activation
Description: Change from week 8 to week 16 in CD4+ T-cell activation, defined as the %CD38+/HLA-DR+
Time Frame: week 8 and week 16
Population: This is an as-treated analysis, limited to 36 subjects who have data for baseline and week 8 and who remain on study treatment through week 8. Among these 36 subjects, 30 subjects with valid data at week 8 and week 16 were included in this secondary analysis.
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 30
percentage | 0.45 [-0.80 to 1.60]

10. Secondary Outcome: Change in CD8+ T-cell Activation
Description: Change from baseline to week 4 in CD8+ T-cell activation, defined as the %CD38+/HLA-DR+, where baseline value is the average of pre-entry and entry
Time Frame: baseline and week 4
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 35
percentage | -0.05 [-4.35 to 3.15]

11. Secondary Outcome: Change in CD8+ T-cell Activation
Description: Change in CD8+ T-cell activation defined as the %CD38+/HLA-DR+ from baseline to week 8, where baseline is the average of pre-entry and entry
Time Frame: Baseline and Week 8
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 33
percentage | -0.450 [-1.75 to 1.95]

12. Secondary Outcome: Change in CD8+ T-cell Activation
Description: Change in CD8+ T-cell activation defined as the %CD38+/HLA-DR+ from week 8 to week 16
Time Frame: week 8 and week 16
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 30
percentage | -0.15 [-1.9 to 6]

13. Secondary Outcome: Change in Proportion of Cycling CD8+
Description: Change from baseline to week 4 in cycling CD8+ , defined as the %Ki67+, where baseline value is the average of pre-entry and entry
Time Frame: baseline and week 4
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 36
percentage | -0.125 [-0.55 to 0.275]

14. Secondary Outcome: Change in Proportion of Cycling CD8+
Description: Change from baseline to week 8 in cycling CD8+ , defined as the %Ki67+, where baseline value is the average of pre-entry and entry
Time Frame: baseline and week 8
Population: This is an as-treated analysis, limited to 36 subjects who have data for baseline and week 8 and who remain on study treatment through week 8. Among these 36 subjects, 32 subjects with valid data at baseline and week 8 were included in this secondary analysis.
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 32
percentage | 0.1 [-0.425 to 0.775]

15. Secondary Outcome: Change in Proportion of Cycling CD8+
Description: Change from week 8 to week 16 in cycling CD8+ , defined as the %Ki67+
Time Frame: from week 8 to week 16
Population: This is an as-treated analysis, limited to 36 subjects who have data for baseline and week 8 and who remain on study treatment through week 8. Among these 36 subjects, 29 subjects with valid data at both week 8 and week 16 were included in this secondary analysis.
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 29
percentage | 0.300 [-0.5 to 0.9]

16. Secondary Outcome: Change in Proportion of Cycling CD4+
Description: Change from baseline to week 4 in cycling CD4+ , defined as the %Ki67+, where baseline value is the average of pre-entry and entry
Time Frame: baseline and week 4
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 36
percentage | 0.125 [-0.375 to 0.575]

17. Secondary Outcome: Change in Proportion of Cycling CD4+
Description: Change from baseline to week 8 in cycling CD4+ , defined as the %Ki67+, where baseline value is the average of pre-entry and entry
Time Frame: baseline and week 8
Population: This is an as-treated analysis, limited to 36 subjects who have data for baseline and week 8 and who remain on study treatment through week 8. Among these 36 subjects, 32 subjects with valid data at both baseline and week 8 were included in this secondary analysis.
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 32
percentage | 0.025 [-0.575 to 0.40]

18. Secondary Outcome: Change in Proportion of Cycling CD4+
Description: Change from week 8 to week 16 in cycling CD4+ , defined as the %Ki67+
Time Frame: week 8 and week 16
Population: as for outcome 15
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 29
percentage | 0.2 [-0.3 to 0.8]

19. Secondary Outcome: Change in Blood Phosphate Levels
Description: Change in blood phosphate levels from baseline to week 4, where baseline value is the average of pre-entry and entry
Time Frame: from baseline to week 4
Population: Among 40 subjects enrolled in A5296, 39 subjects with valid data at both baseline and week 4 were included in this secondary analysis.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 39
mg/dL | 0 [-0.20 to 0.60]

20. Secondary Outcome: Change in Blood Phosphate Levels
Description: Change in blood phosphate levels from baseline to week 8
Time Frame: Baseline to Week 8
Population: Among 40 subjects enrolled in A5296, 37 subjects with valid data at both baseline and week 8 were included in this secondary analysis.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 37
mg/dL | -0.1 [-0.3 to 0.2]

21. Secondary Outcome: Change in Blood Phosphate Levels
Description: Change in blood phosphate levels from week 8 to week 16
Time Frame: from week 8 to week 16
Population: Among 40 subjects enrolled in A5296, 34 subjects with valid data at both week 8 and week 16 were included in this secondary analysis.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 34
mg/dL | 0.10 [-0.30 to 0.40]

22. Secondary Outcome: Change in log10 HIV RNA Levels
Description: Change in log10 HIV RNA levels from baseline to week 4, where baseline value is the average of pre-entry and entry
Time Frame: baseline and week 4
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: log10(copies/mL)
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 36
log10(copies/mL) | 0.02 [-0.09 to 0.14]

23. Secondary Outcome: Change in log10 HIV RNA Levels
Description: Change in log10 HIV RNA levels from baseline to week 8, where baseline value is the average of pre-entry and entry
Time Frame: baseline and week 8
Population: This is an as-treated analysis, limited to 36 subjects who have data for baseline and week 8 and who remain on study treatment through week 8. All 36 subjects had valid data at both baseline and week 8 and were included in this secondary analysis.
Measure: Median (Inter-Quartile Range); unit: log10(copies/mL)
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 36
log10(copies/mL) | -0.02 [-0.12 to 0.10]

24. Secondary Outcome: Change in log10 HIV RNA Levels
Description: Change in log10 HIV RNA levels from week 8 to week 16
Time Frame: week 8 and week 16
Population: This is an as-treated analysis, limited to 36 subjects who have data for baseline and week 8 and who remain on study treatment through week 8. Among these 36 subjects, 34 subjects with valid data at both week 8 and week 16 were included in this secondary analysis.
Measure: Median (Inter-Quartile Range); unit: log10(copies/mL)
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 34
log10(copies/mL) | 0.16 [-0.11 to 0.31]

25. Secondary Outcome: Change in CD4+ T-cell Counts
Description: Change in CD4+ T-cell counts from baseline to week 4, where baseline is the average of pre-entry and entry
Time Frame: baseline and week 4
Population: This is an as-treated analysis, limited to 36 subjects who have data for baseline and week 8 and who remain on study treatment through week 8. Among these 36 subjects, 35 subjects with valid data at both baseline and week 4 were included in this secondary analysis.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 35
cells/mm^3 | -25 [-86 to 40]

26. Secondary Outcome: Change in CD4+ T-cell Counts
Description: Change in CD4+ T-cell counts from baseline to week 8, where baseline is the average of pre-entry and entry
Time Frame: baseline and week 8
Population: This is an as-treated analysis, limited to 36 subjects who have data for baseline and week 8 and who remain on study treatment through week 8. Among these 36 subjects, 36 subjects with valid data at both baseline and week 8 were included in this secondary analysis.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 36
cells/mm^3 | -14 [-70 to 45]

27. Secondary Outcome: Change in CD4+ T-cell Counts
Description: Change in CD4+ T-cell counts from week 8 to week 16
Time Frame: week 8 and week 16
Population: as for outcome 24
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 34
cells/mm^3 | -1 [-93 to 69]

28. Secondary Outcome: Change in IL-6
Description: Changes in levels of systemic inflammation marker IL-6 from baseline to week 4, where baseline is the average of pre-entry and entry
Time Frame: baseline and week 4
Population: This is an as-treated analysis, limited to 36 subjects who have data for baseline and week 8 and who remain on study treatment through week 8. All subjects had valid data at both baseline and week 4 and were included in this secondary analysis.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 36
pg/mL | 0.28 [-0.13 to 0.72]

29. Secondary Outcome: Change in IL-6
Description: Changes in levels of systemic inflammation marker IL-6 from baseline to week 8, where baseline is the average of pre-entry and entry
Time Frame: baseline and week 8
Population: This is an as-treated analysis, limited to 36 subjects who have data for baseline and week 8 and who remain on study treatment through week 8. All 36 subjects with valid data at both baseline and week 8 were included in this secondary analysis.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 36
pg/mL | -0.02 [-0.58 to 0.63]

30. Secondary Outcome: Change in IL-6
Description: Changes in levels of systemic inflammation marker IL-6 from week 8 to week 16
Time Frame: week 8 and week 16
Population: as for outcome 24
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 34
pg/mL | 0.19 [-0.43 to 1.07]

31. Secondary Outcome: Change in C-reactive Protein (CRP)
Description: Changes in levels of systemic inflammation marker CRP from baseline to week 4, where baseline is the average of pre-entry and entry
Time Frame: baseline and week 4
Population: This is an as-treated analysis, limited to 36 subjects who have data for baseline and week 8 and who remain on study treatment through week 8. All 36 subjects with valid data at both baseline and week 4 were included in this secondary analysis.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 36
ng/mL | -141 [-1283.5 to 845]

32. Secondary Outcome: Change in CRP
Description: Changes in levels of systemic inflammation marker CRP from baseline to week 8, where baseline is the average of pre-entry and entry
Time Frame: Baseline and Week 8
Population: as for outcome 29
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 36
ng/mL | 45.5 [-652.5 to 1539.5]

33. Secondary Outcome: Change in CRP
Description: Changes in levels of systemic inflammation marker CRP from week 8 to week 16, where baseline is the average of pre-entry and entry
Time Frame: week 8 and week 16
Population: as for outcome 24
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 34
ng/mL | -34 [-493 to 527]

34. Secondary Outcome: Change in D-dimer
Description: Change in levels of coagulation biomarker d-dimer from baseline to week 4, where baseline value is the average of pre-entry and entry
Time Frame: baseline and week 4
Population: as for outcome 31
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 36
ng/mL | 5.95 [-28.87 to 55.02]

35. Secondary Outcome: Change in D-dimer
Description: Change in levels of coagulation biomarker d-dimer from baseline to week 8, where baseline value is the average of pre-entry and entry
Time Frame: baseline and week 8
Population: as for outcome 29
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 36
ng/mL | 20.30 [-16.08 to 74.90]

36. Secondary Outcome: Change in D-dimer
Description: Change in levels of coagulation biomarker d-dimer from week 8 to week 16
Time Frame: week 8 and week 16
Population: as for outcome 24
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 34
ng/mL | -17.15 [-66.00 to 25.80]

37. Secondary Outcome: Change in Tissue Factor
Description: Change in levels of coagulation biomarker tissue factor from baseline to week 4, where baseline value is the average of pre-entry and entry
Time Frame: baseline and week 4
Population: as for outcome 31
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 36
pg/mL | -2.47 [-6.03 to 0.15]

38. Secondary Outcome: Change in Tissue Factor
Description: Change in levels of coagulation biomarker tissue factor from baseline to week 8, where baseline value is the average of pre-entry and entry
Time Frame: baseline and week 8
Population: This is an as-treated analysis, limited to 36 subjects who have data for baseline and week 8 and who remain on study treatment through week 8. All 36 subjects had valid data at both baseline and week 8 were included in this secondary analysis.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 36
pg/mL | -2 [-6.7 to -0.1]

39. Secondary Outcome: Change in Tissue Factor
Description: Change in levels of coagulation biomarker tissue factor from week 8 to week 16
Time Frame: week 8 and week 16
Population: as for outcome 24
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 34
pg/mL | 3.8 [0 to 8]

40. Secondary Outcome: Change in Total Cholesterol
Description: Change in total cholesterol from baseline to week 8, where baseline value is the average of pre-entry and entry
Time Frame: baseline and week 8
Population: This is an as-treated analysis, limited to 36 subjects who have data for baseline and week 8 and who remain on study treatment through week 8. Among these 36 subjects, 35 subjects with valid data at both baseline and week 8 were included in this secondary analysis.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 35
mg/dL | -12.5 [-28.50 to 5.50]

41. Secondary Outcome: Change in Total Cholesterol
Description: Change in total cholesterol from week 8 to week 16
Time Frame: week 8 and week 16
Population: This is an as-treated analysis, limited to 36 subjects who have data for baseline and week 8 and who remain on study treatment through week 8. Among these 36 subjects, 33 subjects with valid data at both week 8 and week 16 were included in this secondary analysis.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 33
mg/dL | 9 [-4 to 25]

42. Secondary Outcome: Change in LDL Cholesterol
Description: Change in fasting LDL cholesterol from baseline to week 8, where baseline value is the average of pre-entry and entry
Time Frame: baseline and week 8
Population: This is an as-treated analysis, limited to 36 subjects who have data for baseline and week 8 and who remain on study treatment through week 8. Among these 36 subjects, 34 subjects with valid data at both baseline and week 8 were included in this secondary analysis.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 34
mg/dL | -18.25 [-32.20 to 1.50]

43. Secondary Outcome: Change in LDL Cholesterol
Description: Change in fasting LDL cholesterol from week 8 to week 16
Time Frame: week 8 and week 16
Population: This is an as-treated analysis, limited to 36 subjects who have data for baseline and week 8 and who remain on study treatment through week 8. Among these 36 subjects, 32 subjects with valid data at both week 8 and week 16 were included in this secondary analysis.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 32
mg/dL | 14.20 [-0.50 to 32.5]

44. Secondary Outcome: Change in HDL Cholesterol
Description: Change in fasting HDL cholesterol from baseline to week 8, where baseline value is the average of pre-entry and entry
Time Frame: baseline and week 8
Population: as for outcome 40
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 35
mg/dL | 0.50 [-5 to 4]

45. Secondary Outcome: Change in HDL Cholesterol
Description: Change in fasting HDL cholesterol from week 8 to week 16
Time Frame: from week 8 to week 16
Population: as for outcome 41
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 33
mg/dL | 1 [-3 to 5]

46. Secondary Outcome: Change in Non-HDL Cholesterol
Description: Change in non-HDL cholesterol from baseline to week 8, where baseline value is the average of pre-entry and entry
Time Frame: baseline and week 8
Population: as for outcome 40
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 35
mg/dL | -12 [-25 to 2]

47. Secondary Outcome: Change in Non-HDL Cholesterol
Description: Change in non-HDL cholesterol from week 8 to week 16
Time Frame: week 8 and week 16
Population: as for outcome 41
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 33
mg/dL | 4 [-2 to 24]

48. Secondary Outcome: Change in Fasting Glucose
Description: Change in fasting glucose from baseline to week 8, where baseline value is the average of pre-entry and entry
Time Frame: baseline and week 8
Population: as for outcome 23
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 36
mg/dL | -2 [-12.75 to 2.92]

49. Secondary Outcome: Change in Fasting Glucose
Description: Change in fasting glucose from week 8 to week 16
Time Frame: week 8 and week 16
Population: as for outcome 24
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 34
mg/dL | 3.5 [-3 to 15]

50. Secondary Outcome: Primary Adverse Events
Description: Number of subjects experiencing primary adverse events, defined as all reported Grade ≥ 2 signs and symptoms, Grade ≥ 2 laboratory abnormalities and other serious adverse events (SAEs)
Time Frame: baseline and week 16
Population: All 40 subjects enrolled in A5296 were included in this analysis.
Measure: Number; unit: participants
Arm/Group | Sevelamer Carbonate
Number analyzed (Participants) | 40
participants | 28

ADVERSE EVENTS:
Time Frame: AEs reported from study enrollment until study completion at week 16
Description: AE reporting followed DAIDS reporting level
Arm/Group | Sevelamer Carbonate
Serious Adverse Events (participants affected / at risk) | 2/40
Other Adverse Events (participants affected / at risk) | 32/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sevelamer Carbonate (N=40)
Cellulitis (Infections and infestations) | 1
Joint injury (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sevelamer Carbonate (N=40)
Conjunctivitis (Eye disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Alanine aminotransferase increased (Investigations) | 2
Blood bicarbonate decreased (Investigations) | 9
Blood calcium decreased (Investigations) | 8
Blood cholesterol increased (Investigations) | 11
Blood glucose decreased (Investigations) | 5
Blood glucose increased (Investigations) | 9
Blood phosphorus decreased (Investigations) | 10
Blood sodium decreased (Investigations) | 3
Haemoglobin decreased (Investigations) | 2
Low density lipoprotein increased (Investigations) | 6
Neutrophil count decreased (Investigations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No